CLINICAL TRIAL: NCT00879801
Title: Evaluation of Genetic, Biochemical and Clinical Determinants of Type 2 Diabetes Progression in Subjects at High Risk
Brief Title: Genetic Physiopathology and Evolution of Type 2 Diabetes
Acronym: GENFIEV
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: Italian Society of Diabetology (Other); Eli Lilly and Company (Industry)
Responsible Party: FoRiSID, Research Foundation of the Italian Society of Diabetology
Other Study IDs: GENFIEV
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Pre-Diabetes
Keywords: prevention of diabetes; susceptibility genes; type 2 diabetes; insulin resistance; beta-cell funtion
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma sample, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects with IGR: Subjects at high risk of diabetes, such as those with impaired glucose regulation (IFG and or IGT)

SUMMARY:
There are few longitudinal studies in the Caucasian population and even less in the Italian population in subjects with impaired glucose regulation to allow:

1. An estimate of the rate of conversion to type 2 diabetes;
2. To identify subjects at risk; and
3. To assess the physiopathologic mechanisms responsible for the conversion.

In order to set up a longitudinal study capable of defining the above parameters it is mandatory that the physiological, biochemical, and, genetic markers specific for IGR are identified. The goals of the present research proposal are:

1. To clarify the physiological mechanisms responsible for IGR;
2. To identify the biochemical and beta-cell auto-immune parameters present in IGR;
3. Identify genetic markers.

The subjects who will be identified will add up to other 900 individuals who will be recruited as part of a follow-up program sponsored by the Italian Society of Diabetes, specifically designed to assess conversion rate to diabetes.

DETAILED DESCRIPTION:
The main goal of the present research program is to recruit about 600 new subjects with IGR to be added to the 900 subjects which are collected as part of the GENFIEV project which has been designed as a 6-yr follow-up study to ascertain the rate of conversion to type 2 diabetes in the Italian population. In particular the goal of the present research program will be to determine in a sample of the Italian population at greater risk for type 2 diabetes than the general population:

* the pathophysiologic mechanisms responsible for the disorders of impaired glucose regulation (IGR). In particular we will evaluate insulin action and insulin secretion as a function of the degree of glucose tolerance by analyzing these parameters in normal subjects as well as in IFG/NGT, NFG/IGT, and IFG/IGT individuals;
* the biochemical markers associated with the disorders of impaired glucose regulation (IGR). In particular we will evaluate several biochemical parameters (lipid profile, coagulative profile, microlbuminuria, free-fatty acids, PAI-1, fibrinogen, creatinine, uric acid, HbA1c);
* the cardiovascular risk profile associated with the disorders of impaired glucose regulation (IGR). In particular, the relevant biochemical parameters will be integrated with measurements of arterial blood pressure as well as ECG recording;
* the genetic markers associated with the disorders of impaired glucose regulation (IGR). In particular subjects will be screened for HHEX, IGF2,BP2 CDKAL1,TCF2L7, CDKN2A/B,WFS1;
* the impact of environmental factors on the disorders of impaired glucose regulation (IGR).

Finally, we will endeavour to assess the cellular pathways that may be affected by metabolic alterations typically occurring in concomitance with the disorders of impaired glucose regulation (IGR).

ELIGIBILITY:
Inclusion Criteria:

* Each consecutive subject referred to a diabetes clinic for a diagnostic OGTT meeting the above criteria will be assessed as a potential candidate for the study till a total recruitment of 75 individuals will be reached.

  * The OGTT will be performed after an overnight fast as described below.
  * Individuals with IGT (FPG value of < 7.0 mmol/l, and 2-h PG > 7.8 and < 11.1 mmol/l), IFG (FPG > 6.1 and < 7.0 mmol/l, and 2-h PG value of < 11.1 mmol/l).
* Subjects who had both IFG and IGT will included as well.
* Subjects with normal glucose tolerance (FPG <6.1 and 2-h PG <7.8 mmol/l) will be also recruited as controls

Exclusion Criteria:

* Use of drugs known to interfere with glucose metabolism (corticosteroids, beta-blockers, etc)
* Pregnant women, women who are breast feeding
* Active arterial disease (unstable angina, myocardial infarction, cerebrovascular accident, etc) within 3 months of trial entry
* History of malignancy
* Uncontrolled hypertension or hypothyroidism; history of alcohol, or drug abuse, or both
* Active liver disease
* Subjects tacking cyclic hormone replacement therapy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from outpatients diabetic units located in different areas of Italy.
Sampling Method: Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The rate of conversion to diabetes of IGR subjects carrier of type 2 diabetes susceptibility genes | December 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolism, University of Pisa, Pisa, Italy

REFERENCES:
- [Derived] Bianchi C, Miccoli R, Trombetta M, Giorgino F, Frontoni S, Faloia E, Marchesini G, Dolci MA, Cavalot F, Cavallo G, Leonetti F, Bonadonna RC, Del Prato S; GENFIEV Investigators. Elevated 1-hour postload plasma glucose levels identify subjects with normal glucose tolerance but impaired beta-cell function, insulin resistance, and worse cardiovascular risk profile: the GENFIEV study. J Clin Endocrinol Metab. 2013 May;98(5):2100-5. doi: 10.1210/jc.2012-3971. Epub 2013 Mar 28. PMID 23539736